CLINICAL TRIAL: NCT01809951
Title: A Prospective, Open-label, Post-marketing Observational Study to Document the Use of Soy-based Infant Formula With Low Chain Polyunsaturates (LCP) in Infants With Symptoms Suggestive to Cow's Milk Allergy
Brief Title: Isomil Post Marketing Observational Study
Status: Completed | Type: Observational
Sponsor: Melva Louisa (Other)
Responsible Party: Sponsor-Investigator, Melva Louisa, PhD, Indonesia University
Organization: Indonesia University (Other)
Other Study IDs: ANID-1101
Record Dates: First submitted 2013-01-25; First posted 2013-03-13 (Estimated); Last update posted 2017-06-16 (Actual); Status verified 2017-06

CONDITIONS: Cow's Milk Allergy
MeSH Terms: conditions — Milk Hypersensitivity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Isomil Advance with LCP: 4 spoonful of Isomil Advance with LCP in 240 mL of water, 4 times a day

SUMMARY:
The use of soy-isolate protein based formula for infants with cow's milk protein intolerance is common in Indonesia, however, there has not been any systematic collection of clinical data to determine the formula's gastrointestinal tolerance, and the parent's perceptions regarding the formula.

ELIGIBILITY:
Inclusion Criteria:

* infants of 6 - 12 months of age
* full term infants
* birth weight more than 2500 grams
* infants developed symptoms suggestive adverse reactions to cow's milk protein in the investigator's clinical judgements
* subject is prescribed a soy-based infant formula by physician

Exclusion Criteria:

* established/suspected hypersensitivity fo soy
* presence of adverse reactions to cow's milk caused by coincidental infections or other systemic disease
* history of blood group incompatibility, premature delivery, HIV infections, major congenital abnormalities, systemic diseases
* presence of severe gastrointestinal disorder
* subject is participating in any interventional clinical study

Ages: 6 Months to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants with symptoms suggestive adverse reactions to cow's milk protein
Sampling Method: Non-Probability Sample
Enrollment: 534 (Actual)
Dates: Start 2011-08 (Actual); Primary Completion 2013-04 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Parent's acceptance in the feeding of a soy-based infant formula with LCP in infants with symptoms suggestive adverse reactions to cow milk protein | 4-week

SECONDARY OUTCOMES:
percentage of infants with gastrointestinal adverse events | 4-week
percentage of infants with adverse events | 4-week

CONTACTS AND LOCATIONS:
Overall Officials: Zakiudin Munasir, MD, PhD, Principal Investigator — Division of allergy and Immunology, Department of Child Health, Faculty of Medicine, Universitas Indonesia; Sumadiono, MD, PhD, Study Chair — RS Sardjito, Jl Kesehatan No 1 Yogyakarta; Anang Endaryanto, MD, PhD, Study Chair — Allergy Immunology Working Unit, East Java Branch of Indonesian Pediatric Society; Dina Muktiarti, MD, Study Chair — Sub Divisi Alergi Imunologi IKA FKUI, Jakarta; Dewi Kumara Wati, MD, PhD, Study Chair — RSUP Sanglah, Jl Kesehatan No 1-10 Denpasar Bali; Budi Setiabudiawan, MD, PhD, Study Chair — RS Hasan Sadikin Jl Pasteur No 38 Bandung
Locations (1):
- Divisi Alergi Imunologi FKUI RSCM, Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No